CLINICAL TRIAL: NCT01355848
Title: Improving Care Provided to Patients Treated in a Level 1 Trauma Center Post-suicide Attempt
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Stephen O'Connor, Acting Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 39417-C; T32HS013835_1
Record Dates: First submitted 2011-05-10; First posted 2011-05-18 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Suicidal Ideas
Keywords: Suicide; Brief Intervention; Youth; Acute Medical Setting; Readiness to Change; Suicidality
MeSH Terms: conditions — Suicide; Suicidal Ideation | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Intervention (Experimental): The brief intervention consists of stepped care protocol, including building rapport, functional analysis of suicidal behavior, and crisis planning
  Interventions: Behavioral: Brief Intervention for Suicidality
- care as usual (No Intervention): Patients randomized to the care as usual arm will not receive the brief intervention.

INTERVENTIONS:
Behavioral: Brief Intervention for Suicidality — Focuses on behavioral elements of care, including building rapport, functional analysis, and crisis planning
  Arms: Brief Intervention

SUMMARY:
The aim of the study is to refine, elaborate, and pilot a brief intervention for adult patients following a suicide attempt provided during hospitalization in an acute medical setting. 40 participants will be randomized to receive the brief intervention + care as usual or only care as usual. It is hypothesized that the intervention will be acceptable and feasible to both patients and intervention clinicians.

DETAILED DESCRIPTION:
The aim of the study is to refine, elaborate, and pilot a brief intervention for adult patients following a suicide attempt provided during hospitalization in an acute medical setting, and will be addressed with a sample of cases (N = 40) from Harborview. The participants will be randomized into one of two groups: those that receive the intervention and those that do not. All participants will complete a battery of assessments The intervention is based on the theory of teachable moments, wherein timing in proximity to injury and appropriate treatment setting provide a unique opportunity to create patient behavioral change. The brief intervention consists of engaging the patient in conversation regarding suicidal ambivalence (desire to live vs. desire to die), collaborative discovery of primary and secondary drivers of suicidality, and safety planning. A guide to delivering the intervention has been completed and may undergo changes throughout the study. Adherence measures will be developed in order to assess the degree to which the clinician accurately provided the brief intervention without including additional therapeutic elements or leaving out elements required in the intervention guide. Best methods for integrating the brief intervention into services provided on medical and surgical units will be determined, as well.

ELIGIBILITY:
Inclusion Criteria:

* at least 15 years of age
* Inpatient on medical/surgical unit
* Admitted following a suicide attempt
* Sufficient English to benefit from psychotherapy in English
* Consents to be a research participant

Exclusion Criteria:

* Lack of sufficient English to participate in psychotherapy in English
* Prisoner/inmate at time of admission
* Too cognitively impaired, delirious, or psychotic to respond to psychotherapeutic intervention before end of stay on medical/surgical unit. Determination of cognitive impairment, delirium, agitation, and psychosis will be determined through the referral phone call between the PI and the referring care provider, as well as the PI's own clinical assessment of the patient at the outset of the brief intervention.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction Questionnaire | (baseline) Assessment taking place immediately after completion of intervention
  The Patient Satisfaction Questionnaire will be used to determine the acceptability of the intervention by the patient.

SECONDARY OUTCOMES:
Scale for Suicide Ideation | One month follow-up assessment
  The Scale for Suicide Ideation will be used to determine the severity of current suicidality in all participants at the one-month follow-up as compared to the baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen O'Connor, PhD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617